CLINICAL TRIAL: NCT06957730
Title: A Comparison of Hearing Aid Noise Programs on Speech Intelligibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-29404
Record Dates: First submitted 2025-04-22; First posted 2025-05-04 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss, Bilateral or Unilateral
Keywords: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: All participants will be tested with the same three hearing aid programs, but the order of the programs will be randomized for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Phonak Audeo RIC (Experimental): All participants are fit with the Audeo RIC hearing aids, which are programmed with three different settings. All participants are tested with all three settings.
  Interventions: Device: Phonak Audeo Infinio Hearing Aid

INTERVENTIONS:
Device: Phonak Audeo Infinio Hearing Aid — Commercially available receiver-in-canal (RIC) style hearing aid manufactured by Sonova.

SUMMARY:
Hearing impaired participants will be fit with study devices which will have three different hearing aid programs. Speech intelligibility will be measured using validated tests for each of the three hearing aid programs. The order of the hearing aid programs will be randomized across participants and each participant will be blinded as to the programs being tested.

DETAILED DESCRIPTION:
Program 1 is the current default in the commercially available devices. Programs 2 and 3 are being tested against the current default.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral moderate to severe hearing loss (N3-N4)
* Experienced hearing aid user
* Fluent in English
* Cognitively able to complete complex listening tasks

Exclusion Criteria:

* Unilateral hearing loss
* New hearing aid user
* Unable or unwilling to complete complex listening tasks

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
AZBio Speech in noise testing | Day 1 of 1 day study
  A list of 20 sentences is presented from a speaker located in front of the participant. At the same time, background noise is presented from the same speaker at various SNR (Signal to Noise Ratio) levels. That is, speech may be presented 5 dB lower/softer than the noise up to 5 dB higher/louder than the noise. The number of words correct is counted and a percentage from the total number of words presented is calculated. A higher percentage is better and indicates better speech intelligibility. This test will be conducted for all three hearing aid program settings.

SECONDARY OUTCOMES:
Subjective ratings of sound quality | Day 1 of 1 day study
  Participants will be asked to choose between two of the hearing aid programs using an A/B comparison, on the following dimensions: clarity, speech naturalness, speech volume, noise intrusion, listening effort, overall sound quality, and preference. Participants will compare program setting 1 to program setting 2 and choose their preference for each above mentioned dimension. Additionally, participants will compare program setting 1 to program setting 3 and choose preference for each dimension. There is no better or worse, but a count will be taken of preferences for each program. Program 2 and 3 are not compared against each other as the objective of the measure is to compare programs 2 and 3 against the current default program (program 1).

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data collected in this study will only be available to Sonova researchers